CLINICAL TRIAL: NCT00239967
Title: A Randomized, Double-Blind, Two-Arm Placebo-Controlled, Parallel-Group, Multicenter Study of Rimonabant 20 mg Once Daily in the Treatment of Atherogenic Dyslipidemia in Abdominally Obese Patients
Brief Title: An International Study of Rimonabant in Dyslipidemia With AtheroGenic Risk In Abdominally Obese Patients
Acronym: ADAGIO-lipids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC5823
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2009-04-07 (Estimated); Status verified 2009-04

CONDITIONS: Dyslipidemia; Obesity
Keywords: dyslipidemia; obesity
MeSH Terms: conditions — Dyslipidemias; Obesity | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Rimonabant (SR141716)
Drug: Placebo

SUMMARY:
The purpose of this study is to assess the effect of rimonabant 20 mg on HDL (high density lipoprotein) cholesterol and on TG (triglycerides) plasma levels over a period of one year when prescribed with a hypocaloric diet (600 kcal deficit per day) in abdominally obese patients with atherogenic dyslipidemia (low HDL and/or high TG plasma levels). The secondary objectives are to evaluate specific metabolic parameters, visceral fat (in selected sites), safety and tolerability of rimonabant 20 mg.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged >= 18 years
* Waist circumference > 102 cm in men and > 88 cm in women
* Dyslipidemia consisting of:
* Triglyceridemia >= 1.5g/L (i.e. 1.69mmol/L) and ≤ 7.0g/L (i.e. 7.90mmol/L) AND/OR
* HDL cholesterol < 50mg/dL (1.29mmol/L) in women, < 40mg/dL (1.04mmol/L) in men
* If patient with type 2 diabetes are included they must be on a stable dose of oral antidiabetic medication (excluding glitazones) and should not be on insulin therapy
* Written informed consent

Exclusion Criteria:

* Weight change > 5 kg within 3 months prior to screening visit
* Pregnancy or lactation, or women planning to become pregnant
* Absence of medically approved contraceptive methods for females of childbearing potential
* Presence of any other condition (e.g. geographic, social…) actual or anticipated, that the Investigator feels that would restrict or limit the subject's participation for the duration of the study.
* Presence of any clinically significant endocrine disease (other than type 2 diabetes) according to the Investigator
* History of severe depression that could be defined as depression which necessitated the patient to be hospitalized, or patients with 2 or more recurrent episodes of depression or a history of suicide attempt.
* Presence or history of DSM-IV bulimia or anorexia nervosa- Positive test for hepatitis B surface antigen and/or hepatitis C antibody; Abnormal TSH level (TSH > ULN or < LLN ); Hemoglobin < 11g/dL and/or neutrophils > 1,500/mm3 and/or platelets < 100,000/mm3; Positive urine pregnancy test in females of childbearing potential.
* Within 3 months prior to screening visit and between the screening and the inclusion visit:
* Administration of anti obesity drugs (e.g., sibutramine, orlistat)
* Administration of other drugs for weight reduction including herbal preparations (phentermine, amphetamines)
* Thyroid preparations or thyroxine treatment (except in patients on replacement therapy on a stable dose)
* If patients with type 2 diabetes are included they must be on a stable dose of oral antidiabetic medication for at least 3 months and should not be expected to receive insulin therapy within 12 months: Insulin, Glitazones
* Any change in lipid lowering treatment (i.e. introduction of a new drug, change, cessation)- Administration of systemic long-acting corticosteroids- Prolonged use (more than 1 week) of systemic corticosteroids (or if daily dosage > 1000 µg equivalent beclomethasone
* Prolonged administration (more than one week) of antidepressants (including bupropion)
* Prolonged administration (more than one week) of neuroleptics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 803 (Actual)
Dates: Start 2005-05; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
HDL cholesterol and TG plasma levels over a period of one year.

SECONDARY OUTCOMES:
Cholesterol content of HDL2 and HDL3 subfractions,HDL particle size,ApoB,ApoA1,ApoCIII, FFA, indeces of LDL size,hs-CRP,adipokines, fasting glycemia and insulinemia, HbA1c),waist and weight measurements,visceral fat measured by CT scan

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (14):
- Sanofi-aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-aventis Administrative Office, Macquarie Park, Australia
- Sanofi-aventis Administrative Office, São Paulo, Brazil
- Sanofi-aventis Administrative Office, Laval, Canada
- Sanofi-aventis Administrative Office, Hørsholm, Denmark
- Sanofi-aventis Administrative Office, Causeway Bay, Hong Kong
- Sanofi-aventis Administrative Office, Milan, Italy
- Sanofi-aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-aventis Administrative Office, México, Mexico
- Sanofi-aventis Administrative Office, Singapore, Singapore
- Sanofi-aventis Administrative Office, Midrand, South Africa
- Sanofi-aventis Administrative Office, Seoul, South Korea
- Sanofi-aventis Administrative Office, Bromma, Sweden
- Sanofi-aventis Administrative Office, Taipei, Taiwan